CLINICAL TRIAL: NCT04209920
Title: "A Comparison of Two Different Management Techniques for Extensive Molar Defects in Patients Suffering From Molar Incisor Hypomineralization (MIH)" (Randomized Clinical Trial)
Brief Title: A Comparison of Two Different Management Techniques for Extensive Molar Defects in Patients Suffering From MIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hagar Mahmoud Mohie, Teaching Assistant at MSA university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PED 18- 1M
Record Dates: First submitted 2019-09-08; First posted 2019-12-24 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Molar Incisor Hypomineralization; MIH; Hypomineralized; First permanent molar; Molar defects; PMMA; cast adhesive coping
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PMMA crown Group (Active Comparator): Hypomineralized first permanent molars in patients with molar incisor hypomineralization.
  Interventions: Device: CAD-CAM milled PMMA crown
- Cast metal coping Group (Active Comparator): Hypomineralized first permanent molars in patients with molar incisor hypomineralization.
  Interventions: Other: Cast metal coping using nickel chromium alloy

INTERVENTIONS:
Device: CAD-CAM milled PMMA crown — the patient will receive a full coverage restoration for hypomineralized first permanent molar in patient suffering from molar incisor hypomineralization using PMMA disks using a CAD-CAM technology.
  Arms: PMMA crown Group
Other: Cast metal coping using nickel chromium alloy — the patient will receive a full coverage restoration for hypomineralized first permanent molar in patient suffering from molar incisor hypomineralization using Nickel Chromium alloy to make a Cast Coping.
  Arms: Cast metal coping Group

SUMMARY:
It is a randomized clinical trial in which two different types of full coverage restoration in used to restore hypomineralized first permanent molar and protect the remaining tooth structure in patients with molar incisor hypomineralization ,one group is covered with CAD-CAM milled poly methyl methacrylate crowns and the other group is covered with cast metal copings (CAC) using nickel chromium alloy and there will be a nine months follow up.

DETAILED DESCRIPTION:
STUDY POPULATION Sixty (60) hypomineralized molars in patients suffering from molar incisor hypomineralization (MIH) will be randomly selected to share in this study from the out-patient clinic of pedodontics department, Faculty of dentistry, Ain Shams University.

Patient's approval :

All patients and parents will be informed in details about the nature of the investigation and the purpose of the study. They will agree to take part in the study and the parent will sign an informed consent form and the child will have an assent form.

All reasonable steps to protect the security of the personal information and privacy of the patient protected health information will be taken.

All patients will be notice about their privacy practices, their legal duties and their rights.

All patients will be informed about their benefits from research that will be obtaining a restoration to restore and protect the hypomineralized first permanent molars.

Patient's history:

Precise medical, dental and family histories will be taken from all patients through a direct interview and diagnostic sheet.

Parent will be asked about all the possible causes that might cause the molar incisor hypomineralizaion since pregnancy and during the first three years of his life (prenatal, perinatal and postnatal).

Patient's Examination:

* Extra-oral examination: it will be performed following routine procedures to detect any facial abnormality, temporomandibular joint abnormality, any sign of inflammation, pathology or any soft or hard tissue abnormalities.
* Intra oral examination: it will be performed following routine procedures to examine the sound and affected teeth, soft tissue swelling or fistulae, the occlusion and occlusal relation and proximal contacts, the periodontal status and any other anomalies.

Radiographic Evaluation:

Panoramic and peri-apical radiograph for the molar which is indicated to be included on the trial will be taken to the patients preoperatively to evaluate the pulp status, the supporting bone and to ensure that the patients are free from any pathological lesions and to evaluate the position and development of the second permanent molars.

Patient's Grouping:

Selected patients will be randomly divided into two groups:

* Group (I): patients will receive CAD-CAM milled PMMA crown.
* Group (II): patients will receive cast metal coping using nickel chromium alloy.

STUDY PROCEDURE

Clinical steps:

Half of the molars will receive CAD-CAM milled PMMA crown and the other half will receive cast adhesive metal coping using nickel chromium alloy randomly.

1. After proper intraoral and radiographic examination impression of upper and lower arches was made for fabrication of temporary crowns to protect the teeth till fabrication of crowns are finished and the crowns are delivered to the patient.
2. Behavior management of the patient, preparation and administration of local anesthesia is done.
3. Preparation For PMMA crowns Removal of any caries associated to the molar and then reduction of the molar (1mm) all round the molar and (1.5mm) occlusally and impression is taken for upper and lower jaws after reduction for crown fabrication.

   For Cast Adhesive Coping (CAC) Removal of any caries associated to the molar and then reduction of the molar (0.5: 0.7 mm) all round the molar and (1: 1.5mm) occlusally and impression is taken for upper and lower jaws after reduction for crown fabrication.
4. Temporary crown are fabricated and cemented using zinc oxide and eugenol.
5. Delivery and Cementation For PMMA crown After crown is fabricated, the tooth is cleaned, dried and isolated and cementation is done using Self Etch Resin Cement.

   For Cast Adhesive Coping (CAC) After crown is fabricated, the tooth is cleaned and dried and then etched for 30 seconds and then washed and dried to give chalky white appearance, and then the crown is cemented using dual composite cement.
6. Evaluation of quality of both crowns is checked by patient's satisfaction, comfort and function, proper occlusion and proximal contact, margins of the crowns and coverage of all surfaces adequately.
7. The patient will be instructed to maintain good oral hygiene and to avoid eating sticky food.

Then the patient will have 1, 3, 6 and 9 months follow up to evaluate the crowns by clinical examination to evaluate margins and clinical performance of the crowns and gingival hygiene, and bitewing radio graph to evaluate margins of the crowns and any recurrent caries, and questionnaire about related quality of life of the patient to evaluate patient's satisfaction and comfort then data is collected and recorded.

The study is expected to be done in 12 months.

STATISTICAL ANALYSIS A proper statistical method will be carried out to compare between CAD-CAM milled PolyMethyl Methacrylate (PMMA) and Cast adhesive metal coping (CAC) for management of extensive first permanent molar defects in patients suffering from MIH.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with molar incisor hypomineralization having at least one permanent fist molar affected and indicated for full coverage.
2. Patient is healthy and medically free.
3. Patient's age range from 6 to 12 years old.
4. The molar is free from any symptoms of pulp inflammation or has reversible pulpitis (Hypersensitivity).

Exclusion Criteria:

1. Patient who has any chronic systemic disease or immunocompromised.
2. Patient with special health care needs.
3. Molar which has irreversible pulpitis or pulp necrosis.
4. Molar which has periapical radiolucency and/or abscess or fistula or any periapical pathosis.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Marginal Integrity | 9 months follow up
  the crowns is evaluated radiographically using a bite wing radio graph for marginal extension integrity.
Related quality of life: questionnaire | 9 months
  A questionnaire about related quality of life of the patient to evaluate patient's satisfaction and comfort.
Recurrent caries | 9 months
  the tooth is evaluated radiographically using a bite wing radio graph for recurrent caries in the molar.
Gingival Health | 9 months
  the gingival health around the crown is evaluated using Gingival Index (GI) by a periodontal probe and clinical sign of inflammation .
longevity | 9 months
  longevity of the crown is measured by the presence of the crown in the oral cavity cemented and sound.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No